CLINICAL TRIAL: NCT00920504
Title: Pilot Study to Test the Feasibility and the Efficacy of the German Language Adapted PRO-SELF© Plus Pain Control Program, an Educational Intervention Directed at Patients and Their Family Caregivers to Reduce Cancer Pain and Related Symptoms
Brief Title: Pilot Study to Test the Feasibility and the Efficacy of the German Language Adapted PRO-SELF© Plus Pain Control Program
Acronym: PEINCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Basel (Other); University Hospital Freiburg (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PEINCA
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Neoplasm Metastasis
Keywords: Mesh: patient education as topic; Mesh: neoplasms; Mesh: medication therapy management; pain self management; symptom management; education of patients with pain from neoplasm metastases
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- German PRO-SELF(c) Plus PCP (Experimental): Group receives 10 weeks German PRO-SELF(c) Plus PCP intervention program
  Interventions: Behavioral: German PRO-SELF(c) Plus Pain Control Program (PCP)
- Standard Care (Active Comparator): control group receives attention control and standard care
  Interventions: Behavioral: German PRO-SELF(c) Plus Pain Control Program (PCP); Other: Standard Care

INTERVENTIONS:
Behavioral: German PRO-SELF(c) Plus Pain Control Program (PCP) — Educational intervention directed at patients and their family caregivers to reduce cancer pain and related symptoms
Other: Standard Care — Patients in the standard care group will receive routine care provided by their treating physicians without any further care concerning the PRO-SELF© PCP. Patients in the standard care group will be seen by a research nurse in their homes at weeks 1, 2, 4, 6, 8 and 10 and telephone interviews will be conducted at weeks 3, 5, 7 and 9 but the focus of the visits and phone calls will be data collection only.
  Arms: Standard Care

SUMMARY:
The purpose of this pilot study is to refine and test an advanced and adapted German version of the PRO-SELF© Plus Pain Control Program (PCP), an educational intervention directed at cancer pain patients and their families to enhance their pain self management abilities, and to calculate effect sizes for the planning of a sufficiently powered randomized controlled trial (RCT).

DETAILED DESCRIPTION:
Background: Cancer patients experience multiple symptoms throughout the different stages of their illness, with pain as one of the most frequent. Even though effective treatment options exist, more than 40% of all cancer pain patients do not receive adequate pain management. For pain control, in addition to state of the art treatment by professionals, patients and their family caregivers (FCs) have to use self care strategies on a daily basis, a complex process that profits from targeted support by health care providers (HCPs). In phase 1 of this study, the intervention and the study instruments have been translated, adapted and advanced.

Aims: The purpose of this pilot study is to refine and test an advanced and adapted German version of the PRO-SELF© Plus Pain Control Program (PCP), an educational intervention directed at cancer pain patients and their families to enhance their pain self management abilities, and to calculate effect sizes for the planning of a sufficiently powered randomized controlled trial (RCT).

Methods: The advanced and adapted German version of the PRO-SELF© Plus PCP will be tested in a pilot RCT in cancer patients with pain from bone metastasis, compared with standard care, with effect sizes being calculated for the planning of a sufficiently powered RCT. A qualitative sub study will explore patients' and FCs' experiences with pain management, with the educational intervention, and their view of burden and benefit from study participation.

Intervention: The PRO-SELF© Plus PCP is based on three key strategies: (a) provision of information, (b) skill building, and (c) nurse coaching. The 10-week educational program comprises a structured part (teaching of pain management skills including the use of a weekly pillbox, the use of a pain management diary and written instructions on how to communicate with the physician about unrelieved pain) and a tailored part. The patient's answers on questions about his knowledge of pain management serve as basis for tailoring the teaching (academic detailing).

Data analysis: Main outcome variables will be average and worst pain as reported daily by the patient. In order to determine effect sizes for main effect of group, main effect of time and the group by time interaction a repeated measure longitudinal design will be used employing a linear mixed model approach. For the qualitative part, interviews will be analyzed using content analysis.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* with cancer related pain ≥ 3 on a scale of 0-10 during the last two weeks,
* estimated life expectancy of > 6 months as assessed by the physician,
* 18 years of age or older,
* able to understand, read and write German,
* have access to a telephone,
* live in a 1 hour distance around Freiburg or are willing to travel to Freiburg for each visit, agree to participate and give written in-formed consent

Exclusion Criteria:

* documented previous or current psychiatric disorder or cognitive impairment as assessed by the physician (that is, unable to understand and provide informed consent),
* visual or hearing impairment that prevents adequate communication,
* a named FC who is not willing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2009-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
average and worst pain as reported daily by patients on a scale from 0 (no pain) to 10 (worst imaginable pain) | measured daily for 10 weeks and in week 14 and 22

SECONDARY OUTCOMES:
patients' knowledge of cancer pain management | baseline, week 6, 10, 14 and 22

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Spichiger, PhD, Principal Investigator — Institute of Nursing Science, Faculty of Medicine, University of Basel, Switzerland
Locations (1):
- Tumorzentrum Ludwig Heilmeyer Comprehensive Cancer Center Freiburg, Freiburg im Breisgau, Germany

REFERENCES:
- [Derived] Koller A, Miaskowski C, De Geest S, Opitz O, Spichiger E. Results of a randomized controlled pilot study of a self-management intervention for cancer pain. Eur J Oncol Nurs. 2013 Jun;17(3):284-91. doi: 10.1016/j.ejon.2012.08.002. Epub 2012 Sep 4. PMID 22959603
- [Derived] Koller A, Miaskowski C, De Geest S, Opitz O, Spichiger E. Supporting self-management of pain in cancer patients: methods and lessons learned from a randomized controlled pilot study. Eur J Oncol Nurs. 2013 Feb;17(1):1-8. doi: 10.1016/j.ejon.2012.02.006. Epub 2012 Mar 28. PMID 22459260